CLINICAL TRIAL: NCT07045129
Title: Thermal Therapies in the Treatment of Muscle Injuries
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aspetar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F202401070
Record Dates: First submitted 2025-05-22; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Hamstring Injuries; Hamstring Muscle Repair; Hamstring Muscles; Hamstring Rupture; Muscle Tear
Keywords: muscle injury; muscle injuries; hamstring; muscle repair; regeneration; muscle recovery; thermal therapy; CWI; HWI; cold water immersion; hot water immersion; cryotherapy; heat therapy; HD EMG; muscle tear
MeSH Terms: conditions — Hyperthermia | interventions — Cryotherapy; Cold Temperature; Diathermy; Hot Temperature; Rehabilitation

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hamstring injuries grade 1 (Experimental): Grade 1 injury
  Interventions: Other: Cold water immersion; Other: Hot water immersion; Other: Physiotherapy only
- Hamstring injuries grade 2 (Experimental): Grade 2 injury
  Interventions: Other: Cold water immersion; Other: Hot water immersion; Other: Physiotherapy only
- Hamstring injuries grade 3 (Experimental): Grade 3 injury
  Interventions: Other: Cold water immersion; Other: Hot water immersion; Other: Physiotherapy only

INTERVENTIONS:
Other: Cold water immersion — 10 sessions of 15-minute Cold water bath (12°C) after the 10 first physiotherapy sessions.
  Other Names: CWI; cryotherapy; cold
Other: Hot water immersion — 10 sessions of 30 to 45-minute hot water bath (12°C) after the 10 first physiotherapy sessions.
  Other Names: HWI; Heat therapy; hot
Other: Physiotherapy only — Control group. Patients of this group will follow the classic rehabilitation treatment proposed by the physiotherapist and physician of Aspetar without thermal intervention.
  Other Names: rehabilitation

SUMMARY:
Muscle strain injuries represent one of the most prevalent injuries in athletes. Despite this high injury prevalence, there is no evidence to support some of the currently used therapeutic strategies. Amongst them, thermal therapies and especially cryotherapy modalities (Ice, Cold water immersion, perfused garments) have been extensively used on soft tissue injuries to reduce pain perception and decrease inflammation. However, recent findings in humans and in animals have reported conflictual results on the effects of cold on muscle regeneration. On the other hand, recent studies in humans suggest that passive heat exposure can impact positively muscle protein synthesis, mitochondrial content and muscle torque in injured, immobilized and healthy participants. Furthermore, preliminary results from our group have shown a faster removal of muscle damages from the muscle and suggest a better muscle regeneration after a localized heat exposure. As such, our preliminary results confirmed that local heating may represent a promising tool to accelerate muscle regeneration. This randomized controlled trial will investigate the therapeutic effect of two thermal interventions (Hot or cold-water immersion) in the management of acute lower limbs muscle injuries. 135 patients will be distributed in a counterbalanced way into 3 groups: Hot, Cold and Control. All the groups will receive the same physiotherapy treatment. The thermal intervention will consist in 10 sessions of either, 60-minute hot water bath (42°C) for the hot group or, 15-minute Cold water bath (12°C) for the cold group realized after the 10 first physiotherapy session. All thermal interventions will be performed after the testing and physiotherapy treatment.

DETAILED DESCRIPTION:
This randomized controlled trial will evaluate the therapeutic benefits of two different thermal therapies (hot and cold) in the management of lower limb muscle injuries. After meeting the inclusion criteria, participants will be randomized depending on 2 parameters influencing RTS time (injury grading and tendon involvement in the injury) to ensure consistency across groups. The injury will be graded from 0 to 4 using the British athletics muscle injury classification. Participants will follow physiotherapy treatment and receive one of the two thermal therapies or none during the duration of their rehabilitation in Aspetar. Additionally, to the physiotherapy treatment, they will be followed by a researcher to test their evolution on multiple variables during each visit.

First visit to Aspetar:

Patients presenting a potential hamstring injury defined as an acute onset of posterior thigh pain will be examined by a sport physician during their first visit to Aspetar. The procedure detailed succinctly thereafter is part of the clinical routine currently used in Aspetar. To establish a diagnosis, the sport physician will question patient history on the origin, time, intensity, location of his pain and physically examine him. A visual inspection with palpation will be performed where the physician will inspect the presence/absence of ecchymosis and palpate to determine an area of tenderness and pain for the patient. Following the palpation inspection, passive and active flexibility tests will be performed for maximal knee extension and hip flexion with active knee extension. Flexibility will then be assessed using goniometers or inclinometer as the point of maximum tolerable stretch of the hamstring muscle.

The patient will be referred to the radiology department to perform an MRI if the clinical examination indicates a potential hamstring injury defined as:

* Localized pain during palpation of hamstring muscle,
* Increasing pain during isometric contraction,
* Localized pain when performing a passive straight leg test. Before performing the MRI and if the suspected event of the injury was less than 7 days before the visit to Aspetar, the lead PI of the research or a co-investigator will come to the eligible patients to explain them in detail the purpose of this study. If willing to participate in the study, the patient will be invited to read and sign the inform consent form of this study. In case of a non-participation in the study, the patient will be free to continue his rehabilitation treatment in Aspetar. An initial clinical investigation form will be filled with the patient information and injury details.

Based on the MRI results, only patients presenting a confirmed hamstring injury, grade 1, 2 or 3 (BAMIC classification) representing small to extensive tear injuries on one of the following muscles (biceps femoris long head (BFLH), biceps femoris short head (BFSH), semi-membranosus (SM) and semi-tendinosus (ST)) will be included in this study. Grade 0 representing a delayed onset of muscle soreness and considered as MRI-negative for injury and grade 4 injury with a complete muscle tear or tendon avulsion requiring surgery intervention will not be included in this study.

The participant will be asked to signal any supplement and eventual drug or medication consumption. They will also be asked to refrain from taking any drugs and anti-inflammatory particularly non-steroidal anti-inflammatories. Anthropometric characteristics of the patient will be measured before the MRI completion.

Initial and final assessment:

A group of 5 experienced physiotherapists will be selected to treat all the patients included to this study. They will be in charge of performing initial and final assessments for their assigned patients. Initial assessment will be performed during the first physiotherapy session and final assessment will be performed in the 5 days before RTS. They will be blinded to the treatment assigned to the patient. Strength, flexibility, pain perception will be measured during those initial and final assessments. This procedure constitutes the standard rehabilitation procedure of Aspetar.

Randomization procedure:

The participants will be balanced using a Latin square randomization procedure. Following the MR imaging procedure and according to the BAMIC classification, the injuries will be subdivided into 4 grades from 0 to 4. Only injury grades 1, 2 and 3 injuries will be included in the study. Grade 0 and grade 4 injuries will be excluded from this study, but their incidence will be recorded. Injury grading will be the first randomization parameter. The injury location and structure involved (myofascial injury, Musculotendinous junction injury, intra-tendinous injury) will be determined during MRI examination and will be used as a second randomization parameter. Participants will be randomized according to the figure 1. Injury grade and the involvement of tendon in the injury represent two major parameters influencing the time to return to play. To ensure consistency across the 3 interventional group (Hot, Cold and Control), participants will be randomly distributed considering these 2 parameters.

Pre-defined random sequences (using A, B, C sequences, corresponding to the assignment order of the conditions) will be assigned for each of the experiment arms prior to the experiment start. An electronic Latin square generator randomizing the 3 conditions will be used.

Blinding:

The participant will not be blinded on his injury diagnosis and his treatment. It appears impossible to blind the participant on this aspect of the protocol.

The sport medicine physician performing the initial and the return to sport assessment will be blinded to the allocated intervention group, the treatment provided, and the examination performed by the assessor.

The blinded assessor performing the standardized initial and the final RTS clinical examination will be blinded to the assessments of the sports medicine physician, the allocated intervention of the participants and to the radiological diagnosis.

The radiologist scoring the MRIs will be blinded to all clinical information and assessments.

MRI injury detection:

A baseline MRI will be obtained within 7 days of an injury to confirm the presence of a lesion in one of the following muscles and associated tendinous structures: biceps femoris, semimembranosus, semitendinosus. If the participant is included in the study, a second MRI of the injury will be performed in the 5 days preceding the return to sport clearance by the medical team.

MRI will be obtained and processed by Aspetar Radiology department. MRI images will be scored by a senior radiologist from Aspetar radiology department using a standardized scoring form. The BAMIC scale will be used to grade lesion. Only participants with injuries identified by MRI as grade 1, 2 and 3, will be included in the experiment. The standardized scoring form will include the location of the injury (biceps femoris long head (BFLH), biceps femoris short head (BFSH), semimembranosus (SM), semitendinosus (ST)), the injury grade (0, 1, 2, 3, 4), oedema dimensions (craniocaudal length and cross-sectional area), distance of oedema from the ischial tuberosity (to the cranial pole of the oedema and to the highest signal intensity, including intermuscular oedema presence), the presence and extent of intramuscular tendon injury, transverse and mixed connective tissue gap presence, scar morphology, callus gap presence among others.

The participants will be followed-up monthly during the year following their RTS. They will be asked to come back to Aspetar in case of any event with unusual increase of pain or re-injury at the same site than the first injury. After examination of the suspected re-injury by a sport medicine physician, a follow-up MRI of the injury will be performed.

Physiotherapy treatment:

All the participants will perform their rehabilitation treatment in the physiotherapy department of Aspetar. They will follow the Aspetar criteria-based rehabilitation and will be asked to come to Aspetar a minimum of 4 to 6 days a week until return to play clearance. Participants will be cleared for return to sport (RTS) by their treating sports medicine physician if they successfully and asymptomatically complete their criteria-based physiotherapy program and sports-specific (field-based) training. A specialist sports-specific rehabilitator will supervise this last sports-specific phase.

Abbreviated description of the treatment protocol stages, progression and differences.

Thermal interventions:

Participants will be randomly assigned to one of the three following groups: heat, cold, or control without thermal intervention. The physiotherapy treatment will be performed for all participant until their return to sport clearance regardless of their group. The thermal interventions will be performed during a maximum of 10 sessions and realized immediately after the physiotherapy appointments. The thermal intervention will consist in a local heating or cooling using repeated water immersion in a CryoSpa or a ThermoSpa (CET ltd, Northern Ireland). After the 10 first sessions of thermal interventions, the participant will continue his physiotherapy without thermal intervention. Briefly, the lower limbs will be immersed in the corresponding bath, up to the waist to ensure the cooling or heating of the injured area. The participants will be asked to come to Aspetar 4 to 6 days a week to perform their rehabilitation treatment (physiotherapy session + corresponding thermal intervention immediately after each physiotherapy session) until the completion of the rehabilitation protocol and return to play clearance. All thermal interventions will be started as close as possible to the injury detection.

Heat intervention will consist in a 45 to 60-minute bath in a 42 degrees Celsius water following each physiotherapy session. Depending on the participant's tolerance, the bath duration will be modulated during the first visits. A heat acclimation process is expected during the first week of intervention. Cooling solutions (ice, iced towels, cold packs) and cold-water bottles will be provided ad libitum to the participant to limit the core temperature increase and maintain his/her comfort perception high. To assess tolerability and ensure the safety of the participant on the first bath, participants will be given a telemetric core temperature (e-Celsius Performance, Bodycap, France) pill which will indicate in real time their core temperature. Participants will be instructed to swallow the pill with water before their intervention. A second telemetric pill will be given to them on their last thermal intervention to assess the heat acclimation effect of the chronic bathing during their rehabilitation.

The cold intervention will consist in a 15 to 20-minute bath in a 12 degrees Celsius water following each physiotherapy session.

During each bath, participants will be asked to give every 15min their thermal sensation and thermal comfort during the bath intervention.

The control group will have no thermal intervention but will follow the Aspetar criteria-based rehabilitation protocol.

Participants will be asked to refrain from applying any other form of thermal therapies (icing) than what will be assigned to them and avoid applying therapies out of Aspetar.

If a participant completes less than 8 thermal therapy sessions in total, his results will also be censored from the study results.

Return to sport decision:

To be considered able to return to sport the participant will have to meet the criteria for RTS during an assessment by a blinded physiotherapist assessor and an examination by his treating sport medicine physician. The Aspetar decision based RTS model will be used during both of the examinations.

Consensus meetings to agree on RTS dates for every participant will be performed. The following decision algorithm will be used: (1) if the final sports specific training session and discharge by the sports medicine physician is performed on different days, the day of final sports-specific training will be decided as the date of return to sport, (2) if a participant decided to play a game or fully train with their team before discharge, this will noted as the self-decided return to sport and a deviation from protocol, (3) if a participant stop coming (ie, lost to follow-up) or for some reason does not complete the protocol, he will be censored at the latest date he will be seen for physiotherapy (days from injury until last physiotherapy session will be calculated outside of this consensus).

Re-injury follow-up:

Ekstrand et al, (2023) described around 20% of the players experiencing a recurrence of hamstring injury in a UEFA men professional players cohort. A recurrence of the injury is anticipated for a part of the patient during the rehabilitation treatment and the follow-up post RTS. It appears important to monitor the re-injury rate. Participants will be advised to contact the researcher in case of any suspected reinjury. In the meantime, a monthly follow-up will be performed by phone to investigate any possible re-injury a patient could have sustained. If a potential re-injury is detected, the participant will be encouraged to come back to Aspetar for the follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Participant reported a sudden event
* Acute onset pain located on the posterior thigh
* Clinical diagnosis of an acute muscle injury defined as:

Localized pain during palpation of the area, Increasing pain during isometric contraction, Localized pain during specific tests.

* MRI confirmed acute muscle lesion grade 1 - 2 - 3 (Pollock et al., 2014) of hamstring muscles
* Available for physiotherapy treatment 4-5 days a week
* MRI of the injury performed in Aspetar within 7 days from the injury
* Available for follow-up
* Compliant with heat or cold-water immersion

Exclusion Criteria:

* Chronic condition, diabetes, or immune compromised state
* Neurological, cardiovascular, pulmonary, or muscular pathology
* Pacemaker wearer
* Metallic prosthesis
* Skin infection
* Under medication: anti-inflammatory treatment, pain killer drugs, fluoroquinolone antibiotics
* Contraindication to MRI
* Previous verified or suspected lower limb muscle injury for the same leg and the same muscle within the last 6 months
* Chronic lower limb muscle problems on the same muscle
* Grade 0 and 4 muscle injury determined by MRI (Pollock et al., 2014)
* Do not have an intention to return to full sport activity
* Do not want to receive one of the therapies / Noncompliance with heat or cold therapies
* Contraindication to heat
* Do not want to comply with follow-up
* Pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 135 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Time to return to sport in days | From enrollment until return to sport (assessed on average up to 6 weeks)
  The time necessary for the patient to be considered ready to return safely to full level of training in his sport, outside the control of a physiotherapist from the hospital.
  Measure: number of days until the patient is discharged to return to sport (in days).
Isometric hamstring strength | Assessed weekly from the first rehabilitation session after enrolment to the last rehabilitation session before return to sport (assessed on average up to 6 weeks)
  Weekly evolution of the isometric strength of the hamstring muscles using a custom built dynamometer using a strain gauge measuring Force in prone position and pushing the heel against a fixed resistance.
  Measure: Peak Force (in Newtons)
Rate of re-injury | 1 year post-RTS
  The number of re-injury occurence in the year following the injury. Re-injury considered as an hamstrings injury occuring in the same side than the original injury.
  Measure: Every re-injury occurring in the the year following return to sport discharge of the athlete.

SECONDARY OUTCOMES:
Self reported pain perception during injury palpation and physical activity (on a visual arbitrary scale 0-10) | Daily until return to sport (assessed on average up to 6 weeks)
  Pain perceived by the patient during daily palpation and daily rehabilitation exercises.
Muscle activation of each hamstring muscle (% difference activation in comparison the uninjured leg) as measured by High Density Electromyography. Determining the amplitude of the EMG signal, conduction velocity and motor units recruitment patterns | Weekly until return to sport (assessed on average up to 6 weeks)
  Muscle activation measured using high density electromyography
Mediolateral width and anterior/posterior depth of the total injured area (in mm) | Study inclusion/return to sport (assessed on average up to 6 weeks)
  Area of the injured site (region of interest) identified on the MRI scan and Ultrasound Scan. Comparison between early and late MRI and US performed during the intervention phase.
Hamstring range of motion using MHFAKE measure (in degrees) | Daily until return to sport (assessed on average up to 6 weeks)
  The MHFAKE (maximal hip flexion Active knee Extension) is performed with the patient supine with hip flexed and actively extending the knee until pain tolerance allows. The maximum knee extension angle is measured with a goniometer to assess hamstrings flexibility.

CONTACTS AND LOCATIONS:
Locations (1):
- Aspetar Orthopaedic and Sports Medicine Hospital, Doha, Qatar

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] D'Souza RF, Figueiredo VC, Markworth JF, Zeng N, Hedges CP, Roberts LA, Raastad T, Coombes JS, Peake JM, Mitchell CJ, Cameron-Smith D. Cold water immersion in recovery following a single bout resistance exercise suppresses mechanisms of miRNA nuclear export and maturation. Physiol Rep. 2023 Aug;11(15):e15784. doi: 10.14814/phy2.15784. PMID 37549955
- [Background] Roberts LA, Raastad T, Markworth JF, Figueiredo VC, Egner IM, Shield A, Cameron-Smith D, Coombes JS, Peake JM. Post-exercise cold water immersion attenuates acute anabolic signalling and long-term adaptations in muscle to strength training. J Physiol. 2015 Sep 15;593(18):4285-301. doi: 10.1113/JP270570. Epub 2015 Aug 13. PMID 26174323
- [Background] Peake JM, Roberts LA, Figueiredo VC, Egner I, Krog S, Aas SN, Suzuki K, Markworth JF, Coombes JS, Cameron-Smith D, Raastad T. The effects of cold water immersion and active recovery on inflammation and cell stress responses in human skeletal muscle after resistance exercise. J Physiol. 2017 Feb 1;595(3):695-711. doi: 10.1113/JP272881. Epub 2016 Nov 13. PMID 27704555
- [Background] McGorm H, Roberts LA, Coombes JS, Peake JM. Turning Up the Heat: An Evaluation of the Evidence for Heating to Promote Exercise Recovery, Muscle Rehabilitation and Adaptation. Sports Med. 2018 Jun;48(6):1311-1328. doi: 10.1007/s40279-018-0876-6. PMID 29470824
- [Background] Hafen PS, Abbott K, Bowden J, Lopiano R, Hancock CR, Hyldahl RD. Daily heat treatment maintains mitochondrial function and attenuates atrophy in human skeletal muscle subjected to immobilization. J Appl Physiol (1985). 2019 Jul 1;127(1):47-57. doi: 10.1152/japplphysiol.01098.2018. Epub 2019 May 2. PMID 31046520
- [Background] Nagata I, Kawashima M, Miyazaki A, Miyoshi M, Sakuraya T, Sonomura T, Oyanagi E, Yano H, Arakawa T. Icing after skeletal muscle injury with necrosis in a small fraction of myofibers limits inducible nitric oxide synthase-expressing macrophage invasion and facilitates muscle regeneration. Am J Physiol Regul Integr Comp Physiol. 2023 Apr 1;324(4):R574-R588. doi: 10.1152/ajpregu.00258.2022. Epub 2023 Mar 6. PMID 36878487
- [Background] Benoit S, Nicolas B, Gregoire MP, Francois B, Abdellah H, Hicham M, Said A, Guillaume C. Hot But Not Cold Water Immersion Mitigates the Decline in Rate of Force Development Following Exercise-Induced Muscle Damage. Med Sci Sports Exerc. 2024 Dec 1;56(12):2362-2371. doi: 10.1249/MSS.0000000000003513. Epub 2024 Jul 4. English, French. PMID 38967392
- [Background] Kawashima M, Kawanishi N, Tominaga T, Suzuki K, Miyazaki A, Nagata I, Miyoshi M, Miyakawa M, Sakuraya T, Sonomura T, Arakawa T. Icing after eccentric contraction-induced muscle damage perturbs the disappearance of necrotic muscle fibers and phenotypic dynamics of macrophages in mice. J Appl Physiol (1985). 2021 May 1;130(5):1410-1420. doi: 10.1152/japplphysiol.01069.2020. Epub 2021 Mar 25. PMID 33764172